CLINICAL TRIAL: NCT04421053
Title: Gestational Weight Gain (GWG) Recommendations for Chinese Women With Gestational Diabetes Mellitus (GDM)
Brief Title: Weight Gain Recommendations for Chinese Women With Gestational Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JS-2333
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-05

CONDITIONS: Gestational Diabetes; Gestational Weight Gain
Keywords: gestational diabetes mellitus; gestational weight gain; blood glucoes monitoring; health management; moblie health
MeSH Terms: conditions — Diabetes, Gestational; Gestational Weight Gain | interventions — Prenatal Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples and stool samples are collected from participants in Beijing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women with GDM: After participants enrollment, we conducted follow-up visit every two weeks. Blood glucose values, body weight, life style record and clinical information are collected. Blood samples and stool samples are collected from participants in Beijing.
  Interventions: Behavioral: prenatal care for women with GDM

INTERVENTIONS:
Behavioral: prenatal care for women with GDM — we conduct prenatal care for GDM pregnancies through both prenatal clinic and app.

SUMMARY:
The 2009 IOM recommendation value for weight gain during pregnancy is widely used. Due to the unclear relationship between gestational diabetes mellitus and weight gain during pregnancy when formulating this recommendation value, pregnant women with gestational diabetes mellitus were excluded from the study population. Control of appropriate weight gain and control of blood glucose stability is an important part of GDM management in pregnant women. The incidence of GDM in China is about 15%-20%, and the number of pregnant women with GDM ranks first in the world. For the sake of the current and long-term health of maternal and infant, it is of great significance to explore the appropriate weight gain range and formulate the recommended value for GDM pregnant women as an independent population. This project intends to use prospective cohort study of combining the observation of pregnant women with gestational diabetes blood sugar and weight changes, through the comparison of normal pregnant women suitable scope of weight gain, analyzes its influence on adverse pregnancy outcomes, increased the weight of gestational diabetes women recommended value is put forward, and combined with the Delphi expert consultation method for evaluation.

DETAILED DESCRIPTION:
This project is a prospective cohort study designed to investigated the changes in blood glucose and body weight in women with gestational diabetes during pregnancy. The study aimed to enroll 4000 participants, using health management app in addition to routine prenatal care. Researchers screen subjects strictly according to the exclusion and inclusion criteria and those who interested sign the informed consent. participants completed baseline questionnaire and dietary questionnaire at app under the instruction of researchers. Pregnant women come back for follow up-visit every 2 weeks until delivery. If anyone doesn't upload the weight data for a week and doesn't respond to the phone call from the researchers, she will be regarded as lost follow-up,the number of lost follow-up cases are supplemented by increasing the enrollment. Data analysis and result output finally.

Besides, part of the study conducted in Beijing has some special points which don't exsit in large cohort study: participants equipment dynamic blood glucose monitor for glycemic control and their blood samples and stool samples will be collected at 24-28, 32 and 36 gestational weeks,respectively.

Based on the description of weight gain range of pregnant women with normal blood glucose, the influence of weight gain on adverse pregnancy outcome was analyzed, and the recommended weight gain value for women with gestational diabetes was proposed in combination with Delphi expert consultation method.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who have regular labor inspection and delivery in the labor inspection hospital;
* Pregnant women with gestational diabetes diagnosed by OGTT at 24 to 28 weeks of pregnancy;
* Singleton pregnancy;
* Those who can skillfully use mobile phones and other electronic devices for scientific follow-up and voluntarily record their daily weight;
* Voluntary signing of informed consent.

Exclusion Criteria:

* Patients with pre-pregnancy diabetes mellitus or abnormal OGTT screening in early pregnancy;
* diabetic ketoacidosis,high blood sugar of high permeability anemia,leukemia, and lymphoma without clinical control.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnancies with gestational diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 4050 (Estimated)
Dates: Start 2020-03-24 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of pregnancy outcomes | delivery
  pregnancy outcomes including preeclampsia, gestational hypertension.
The incidence rate of infant outcomes | delivery
  infant outcomes including SGA,neonatal hypoglycemia.

SECONDARY OUTCOMES:
the value of gestational weight gain during third trimester | from enrollment to delivery
  pregnant women with diabetes mellitus type 2,children with hypertension,obesity,diabetes,cardiovascular disease,etc.

CONTACTS AND LOCATIONS:
Overall Officials: Liangkun Ma, Study Chair — Chinese Academy of Medical Science & Peking Union Medical College Hospital
Locations (1):
- Department of ob gyn, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided